CLINICAL TRIAL: NCT07358364
Title: Remibrutinib in Real-world Clinical Practice: a Prospective, Multi-country, Non-interventional, Effectiveness and Safety Study
Brief Title: Remibrutinib in Real-world Clinical Practice
Acronym: REASSERT
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLOU064A2402
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Remibrutinib; Non-Interventional Study; Chronic Spontaneous Urticaria; Second-generation H1 antihistamine
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Cohort 1: Inadequate control of CSU despite licensed dose of sgH1-AH (no other pre-treatments permitted) and decision to escalate sgH1-AH treatment
- Cohort 2: Inadequate control of CSU despite licensed dose or escalated sgH1-AH(s) (no other pre-treatment with exception of first generation H1-AH permitted) with decision to switch to remibrutinib treatment as per local label
- Cohort 3: Any other treatment received in addition to H1-AH, any time during patients' CSU treatment history, with decision to switch to remibrutinib treatment as per local label

SUMMARY:
Prospective, multi-country, non-interventional study in patients with CSU where the treatment decision prior enrolment has been made to either escalate current sgH1-AHs treatment or escalate/switch current treatment to remibrutinib. The primary aim of this study is to gather real-world effectiveness and safety data for remibrutinib, a new treatment option, covering a broader, real-world clinical practice population.

DETAILED DESCRIPTION:
This is a prospective, multi-country, non-interventional study in patients with CSU where the treatment decision prior enrolment has been made to either escalate current sgH1-AHs treatment or escalate/switch current treatment to remibrutinib. The primary aim of this study is to gather real-world effectiveness and safety data for remibrutinib, covering a broader, real-world clinical practice population. The study employs an umbrella design which brings the evidence needs from multiple countries under the REASSERT global program. Countries will generate local protocol to be used in their country; the local study documentation will be a minimised version of the global document, modified to align with country's evidence needs, given local disparities in treatment guidelines, access, physician type and ePROs/eDiaries used. To achieve the core objectives the observation needs to include either the Urticaria Control Test (UCT) or Urticaria Activity Score over 7 days (UAS7) and the Dermatology Life Quality Index (DLQI). Data from all countries will be pooled and analyzed globally. In certain instances, some modifications of the global protocol may be permitted. For example, in countries where prospective monitoring of off-label antihistamines is prohibited, cohort 1 will not be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of primary CSU by the treating physician.
* Aged at least 18 years on the date of enrolment.
* Written informed consent of the patient to participate in the study (according to country specifications) and willingness to complete full follow-up period of 24 months.
* Cohort-specific observational inclusion criteria:

  * Cohort 1: Inadequate control of CSU despite licensed dose of sgH1-AH (no other pre-treatments permitted) and decision (independent of study enrolment) to escalate sgH1-AH treatment.
  * Cohort 2: Inadequate control of CSU despite licensed dose or escalated sgH1-AH(s) (no other pre-treatment with exception of first generation H1-AH permitted) with decision (independent of study enrolment) to switch to remibrutinib treatment as per local label.
  * Cohort 3: Any other treatment received in addition to H1-AH, any time during patients' CSU treatment history, with decision (independent of study enrolment) to switch to remibrutinib treatment as per local label. Note, occasional steroid rescue medication is out of scope for cohort definition. If a patient had been on continuous steroids for at least three weeks during treatment history, they will be included in cohort 3.

Note: Candidate patients must not have initiated the next escalated treatment step (i.e. up dosed AH for cohort 1, or remibrutinib for cohorts 2 and 3) prior to their enrolment to ensure the baseline visit captures their clinical status before treatment escalation.

Exclusion Criteria:

* Currently enrolled in a clinical trial or on any experimental treatment.
* Patients within the safety follow-up phase of a previous interventional or non-interventional study.
* Patients who received remibrutinib as an investigational medical product during a remibrutinib interventional study or MAP/PSDS at any time in the past.
* Patients not capable or willing to continuously provide ePRO/eDiary data via electronic means throughout the duration of the study.
* Patients who are treated with remibrutinib outside of the local label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CSU where the treatment decision prior enrolment has been made to either escalate current sgH1-AHs treatment or escalate/switch current treatment to remibrutinib
Sampling Method: Non-Probability Sample
Enrollment: 3280 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2031-10-30 (Estimated); Study Completion 2031-10-30 (Estimated)

PRIMARY OUTCOMES:
UCT7 score | 12 weeks after initiating remibrutinib treatment
  Urticaria Control Test is looking retrospectively for 7 days (UCT7) and consists of 4 questions. Each question is scored 0-4, with a total score range of 0 (poor control) to 16 (well controlled).
UAS7 score | 12 weeks after initiating remibrutinib treatment
  Urticaria Activity Score over 7 days UAS7 is based on 2 daily questions scored 0-3 per day, ranging from 0 (complete control) to 42 (poor control)

SECONDARY OUTCOMES:
Number and proportion of participants with well-controlled disease and complete disease | Up to 24 months
  Proportion of patients with UCT score ≥12 and UAS7 score ≤6. Urticaria Control Test (UCT) consists of 4 questions scored 0 (very much) to 4 (not at all), with a total score range of 0 to 16. High scores indicates better disease control. Urticaria Activity Score over 7 days (UAS7) is based on 2 daily questions, with daily score of 0 to 6 and weekly score of 0 to 42. Lower scores suggests urticaria free and well controlled urticaria.
Change from baseline (CFB) in UCT score | Up to 24 months
  Change in UCT score over time. Urticaria Control Test (UCT) consists of 4 questions scored 0 (very much) to 4 (not at all), with a total score range of 0 to 16. Highest scores indicates better disease control. The study is not powered to detect any specific difference and the purpose is to estimate any observed difference descriptively.
Change from Baseline in UAS7 score ≥ minimal important difference | Up to 24 months
  Urticaria Activity Score over 7 days (UAS7) is based on 2 daily questions, with daily score of 0 to 6 and weekly score of 0 to 42. Lower scores suggests urticaria free and well controlled urticaria. The study is not powered to detect any specific difference and the purpose is to estimate any observed difference descriptively.
Change in angioedema activity score (AAS7) from baseline | Up to 24 months
  Angioedema Activity Score (AAS7) is assessing disease activity over 7 days in patients with urticaria. The score is based on 5 daily questions scored 0 (no discomfort) to 3 (severe discomfort), with weekly score ranging from 0 to 15. Higher scores indicates greater severity of angioedema.
Number of weeks without angioedema | Up to 24 months
  Number of weeks without angioedema evaluated using AECT and/or application entries. Angioedema Control Test (AECT) consists of 4 questions evaluating swelling, rated from 0 (not at all) to 4 (very often) with a maximum score of 16, higher score indicating better control.
Number of participants with rescue medication requirement | Up to 24 months
  Number of participants with rescue medication requirement
Characterize CSU relapse | Up to 24 months
  CSU relapse by frequency and presentation
UCT score | Up to 24 months
  Urticaria Control Test (UCT) consists of 4 questions scored 0 (very much) to 4 (not at all), with a total score range of 0 to 16. High scores indicates better disease control. The study is not powered to detect any specific difference and the purpose is to estimate any observed difference descriptively.
UAS7 score | Up to 24 months
  Urticaria Activity Score over 7 days (UAS7) is based on 2 daily questions, with daily score of 0 to 6 and weekly score of 0 to 42. Lower scores suggests urticaria free and well controlled urticaria. The study is not powered to detect any specific difference, descriptive analysis of difference over time will be presented.
Change in AECT from baseline | Up to 12 weeks
  Change in AECT score over time will be presented. The study is not powered to detect any specific difference, descriptive analysis of difference over time will be presented. Angioedema Control Test (AECT) is a 4 item questionnaire evaluating swelling within last 4 weeks. Each question is scored from 0 (not at all) to 4 (never), total score ranging from 0 to16. Higher scores represent a well controlled disease.
Number of participants with administration of remibrutinib as monotherapy | Up to 24 months
  Number of participants with remibrutinib as monotherapy in cohort 2 and 3
Monotherapy duration | Up to 24 months
  Duration of remibrutinib as monotherapy expressed by days, weeks or months in cohort 2 and 3
Number of participants with Administration of remibrutinib as monotherapy with "on demand" sgH1-AH | Up to 24 months
  Number of participants with Administration of remibrutinib as monotherapy with "on demand" sgH1-AH in cohort 2 and 3
Duration of monotherapy with "on demand" sgH1-AH | Up to 24 months
  Duration of remibrutinib therapy with "on demand" sgH1-AH expressed by days, weeks or months in cohort 2 and 3
Number of participants with usage of concomitant sgH1-AHs and additional prescribed CSU treatments | Up to 24 months
  Descriptive analysis of concomitant sgH1-AHs
Number of participants with administration of CSU-related treatment(s) outside of local and/or international guidelines | Up to 24 months
  Number of participants with administration of CSU-related treatment(s) outside of local and/or international guidelines
Demonstrate relationship between non-adherence to local/international guidelines and impact on patient, disease control, treatment patterns and HCRU during early and long-term follow-up | Up to 24 months
  Demonstrate relationship between non-adherence to local/international guidelines and impact on patient, disease control, treatment patterns and HCRU during early and long-term follow-up
Delay of treatment escalation contrary to local and/or international guidelines when UCT <12 or UAS>6 | Up to 24 months
  Delay of treatment escalation contrary within 2-4 weeks from up-dosed sgH1-AH when UCT <12 or UAS>6 at time points measuring UCT7 (early) / UCT (month 3 onwards) / UAS7 group.
  This will be measured by time in days/months without escalation, with UCT<12 or UAS7>6 at time points measuring UCT7 / UCT (month 3 onwards) / UAS7 group
Time without escalation, with UCT<12 or UAS7>6 | Up to 24 months
  Time in days/months without escalation while UCT score is below 12 OR UAS7 score above 6. Urticaria Control Test consists of 4 questions, score below 12 indicates poor disease control. Urticaria Activity Score over 7 days is based on 2 daily questions with a maximum daily score of 6 and weekly total score up to 42. Lower scores indicates better urticaria control.
Number of participants with escalation to remibrutinib | Up to 24 months
  Number of patients with escalation to remibrutinib (cohort 1), time to escalate, prior medications/escalations, and disease control at time of escalation will be presented.
Number of participants with administration of above the licensed dose of sgH1-AH prior to remibrutinib switch | Up to 24 months
  Number of participants receiving escalated doses of sgH1-AH above the licensed dose (2 times, 3 times, 4 times, >4 times) prior to remibrutinib switch. This will be presented for cohort 1 and 2.
Number of sgH1-AH treatment escalations and switches prior to remibrutinib escalation | Up to 24 months
  Number of sgH1-AH treatment escalations and switches prior to remibrutinib escalation
Demonstrate benefit of early vs late treatment escalation to remibrutinib | Up to 24 months
  Demonstrate benefit of early vs late treatment escalation to remibrutinib
Proportion of patients with uncontrolled angioedema escalated to remibrutinib | Up to 24 months
  Presence of angioedema will be reported through App and/or derived from AAS and AECT scores
Proportion of patients requiring corticosteroids prior to switch to remibrutinib | Up to 24 months
  Proportion of patients requiring corticosteroids for disease control prior to switch to remibrutinib (cohort 1 and 2)
Quality of life measured through DLQI score | Up to 24 months
  Dermatology Life Quality Index (DLQI) score consists of 10 questions scored from 0 (no impact at all) to 3 (very much). Total score ranges from 0 to 30, with lower scores showing lowest impact of disease on quality of life.
Quality of life evaluated through Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL) questionnaire scores | Up to 24 months
  Change over time in Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL) questionnaire. CU-Q2oL consists of 20 items rated from 0 (never) to 5 (very often). Total score ranges from 0 to 25, with lower scores showing better urticaria control. The study is not powered to detect any specific difference, descriptive analysis of difference over time will be presented.
Quality of life measured through Sleep interference score | Up to week 12
  Sleep interference will be evaluated though bespoke question. Maximum score along 7 days ranges from 0 to 21, lower scores showing lowest interference of CSU with sleep.
Quality of life measured through Hospital anxiety and depression scale (HADS) | Up to 24 months
  Quality of life will be evaluated through HADS measuring anxiety and depression components, as well as change from baseline in HADS score. Hospital Anxiety and Depression Score (HADS) is a 14 item questionnaire, 7 item rating anxiety and 7 depression. Responses are rated from 0 (never) to 3 (almost all time) at each question. Total score for anxiety and total score for depression range from 0 to 21, higher scores showing higher anxious/depressive symptomatology. Descriptive analysis will be presented.
Number of events related to CSU or Health Care Resource utilisation | Up to 24 months
  Health Care resource utilisation (HCRU) will be evaluated based on quarterly and annualized number of health care resource utilisation related to CSU.
Work productivity and activity impairment (WPAI-CU) score | Up to 24 months
  Work productivity assessed through WPAI questionnaire which consists of 6 questions, used to calculate 4 types of scores, absenteeism (work time missed), presenteeism (impairment at work/reduced on the job effectiveness), work productivity loss (overall work impairment), and activity impairment. The scores are expressed in percentage with higher numbers indicating greater impairment and less productivity at work.
Incidence of AEs | Up to 24 months
  Incidence of AEs, including serious AEs in patients who initiated remibrutinib and in patients with sgH1-AH treatment alone

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Cleaver Dermatology, Kirksville, Missouri, United States

IPD SHARING:
Plan to Share IPD: No